CLINICAL TRIAL: NCT03650283
Title: The Relation Between PRST Score, Skin Conductance and BIS Values During Anesthesia
Brief Title: Relation Between PRST Score, Skin Conductance and BIS
Acronym: RB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bahar SAKIZCI UYAR, MD, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 40/19
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Awakeness, Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: monitoring — The bispectral index (BIS) and skin conductance (SC) monitors will be connected when patient will be positioned on the operating table. A BIS value greater than 60 will be considered an indicator of light anaesthesia. The SC monitoring will be achieved using the MEDSTORM AS 2005 monitor. Number of fluctuations in mean skin conductance (NFSC) of >0.1 s-1 in a period of 15 s might be counted as a significant change and indicates an increase in the sympathetic outflow. General anaesthesia will be performed and laryngeal mask will be inserted. Blood pressure, heart rate, BIS, SC, and PRST (pressure, rate, sweating, tears) score will be recorded.

SUMMARY:
Determine the relation between PRST (pressure, rate, sweating, tears) score, skin conductance (SC) and Bispectral index (BIS) values during anesthesia

DETAILED DESCRIPTION:
Probability of >0 points in the PRST as a function of BIS and number of fluctuations in mean skin conductance (NFSC) will be recorded during the anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Minor elective surgery
* General anaesthesia

Exclusion Criteria:

* autonomic neuropathy
* presence of a pacemaker
* medication with anticholinergic drugs
* use of ketamine, clonidine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-04 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between NFSC, PRST and BIS | anesthesia induction (while giving induction agent to the patient), surgical incision (when the surgeon makes the first incision), extubation (when LMA is removed)
  Correlation between NFSC-PRST and, BIS-PRST will be assessed.